CLINICAL TRIAL: NCT05381662
Title: CD19 Chimeric Antigen Receptors and CD19 Positive Feeder T Cells as a Leukemia Consolidation Treatment
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCT19-T19 v1.1
Record Dates: First submitted 2018-08-05; First posted 2022-05-19 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2022-12

CONDITIONS: Acute Lymphoblastic Leukemia in Remission

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): This cohort will determine the safety and efficacy of CD19 CAR-T cells and CD19 positive feeder T cells for CD19+ acute lymphoblastic leukemia without Chemotherapy pretreatment
  Interventions: Biological: CD19 CAR-T cells and CD19 positive feeder T cells
- Cohort 2 (Experimental): This cohort will determine the safety and efficacy of CD19 CAR-T cells and CD19 positive feeder T cells for CD19+ acute lymphoblastic leukemia with Chemotherapy pretreatment
  Interventions: Biological: CD19 CAR-T cells and CD19 positive feeder T cells

INTERVENTIONS:
Biological: CD19 CAR-T cells and CD19 positive feeder T cells — Detailed Description: Patients were divided into two groups, group 1 and group 2, and each group was enrolled in 5 patients. Group 1 patients did not receive any pretreatment, and group 2 patients received pretreatment with cyclophosphamide and fludarabine prior to reinfusion. Then Patients were given Chimeric Antigen Receptor T-Cell ( CAR-T) and CD19-positive T cells.

SUMMARY:
This is a single center,randomized ,two-cohorts, open-label ,phase 1/2 study to evaluate the efficacy and safety of T cells expressing CD19 chimeric antigen receptors combined with CD19 positive feeder T cells treatment for CD19+ acute lymphoblastic leukemia patients in remission .

DETAILED DESCRIPTION:
Patients were divided into two groups, group 1 and group 2, and each group was enrolled in 5 patients. Group 1 patients did not receive any pretreatment, and group 2 patients received pretreatment with cyclophosphamide and fludarabine prior to reinfusion. Then Patients were given Chimeric Antigen Receptor T-Cell( CAR-T) and CD19-positive T cells.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65
2. Voluntary informed consent is given
3. Expected survival ≥12 weeks
4. Relieve CD19+ acute leukemia
5. Organ function: (1)Left ventricular ejection fractions≥ 0.6 by echocardiography (2)ALT ≤3 times of ULN, or bilirubin <2.0 mg/dl (3)Creatinine < 2 mg/dl and less than 2.5 × normal for age (4)Prothrombin time and activated partial thromboplastin time < 2 times of ULN (5)Arterial oxygen saturation> 92%
6. Karnofsky score ≥ 60 ;
7. No history of combined chemotherapy in the recent 1 month and no immunotherapy in the recent 3 months;

Exclusion Criteria:

1. Uncontrolled active infections
2. Active hepatitis B or hepatitis C infection
3. HIV infection
4. History of myocardio infarction in the past 6 months, or history of severe arrhythmia
5. Congenital immunodeficiency
6. Pregnant or lactating women
7. History or presence of clinically relevant CNS pathology such as epilepsy, generalized seizure disorder, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis
8. Previous treatment with any gene therapy products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-08-02 (Actual); Primary Completion 2024-08-02 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe CRS | 12 months
  The safety of the CD19 CAR-T cells and CD19 positive feeder T cells treatment will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, Ph.D, Study Chair — The First Affiliated Hospital of Soochow University
Locations (2):
- China (2):
  - The first affiliated hospital of soochow university, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou